CLINICAL TRIAL: NCT00064415
Title: A Multicenter, Open-Label, Randomized, Active-Controlled, Parallel Group Chronic Safety Study of (R,R)-Formoterol in the Treatment of Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: To Evaluate the Long-term Safety of (R,R)-Formoterol in Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091-060
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arformoterol tartrate 50 mcg QD
  Interventions: Drug: arformoterol
- 2 (Active Comparator): Salmeterol 42 mcg BID
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: arformoterol — Arformoterol inhalation solution, 50 mcg QD
  Other Names: Brovana Inhalation Solution; (R,R)-Formoterol
  Arms: 1
Drug: Salmeterol — Salmeterol MDI, 42 mcg BID
  Other Names: Serevent MDI; racemic formoterol
  Arms: 2

SUMMARY:
The purpose of this study is to determine the long-term safety of arformoterol over a period of 12 months in subjects with COPD

DETAILED DESCRIPTION:
This was a multicenter, open-label, randomized, active controlled, parallel group chronic safety study of arformoterol 50 mcg once daily over a period of 12 months in subjects with COPD. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
INCLUSION CRITERIA: In order to qualify for participation, subjects must meet the following criteria:

* Must give written informed consent prior to participation. Women of childbearing potential must also sign the Women of Childbearing Potential Addendum.
* Must be willing to comply with study procedures and visit schedule
* Male or female >35 years of age
* Female subjects <65 years of age must have a serum pregnancy test conducted at Visit 1 and confirmed negative prior to randomization. Subjects of childbearing potential must be using an acceptable method of birth control.
* Female subjects who are considered not of childbearing potential must be: (1) documented surgically sterile, OR (2) postmenopausal
* Have a primary diagnosis of COPD, which may include components of chronic bronchitis and/or emphysema. Diagnosis can be made during the screening process.
* Have a minimum smoking history of 15 pack-years (pack-years = the number of cigarette packs per day times the number of years)
* Medical Research Council (MRC) Dyspnea Scale Score >2
* Have a baseline FEV1 <65% of predicted normal value and >0.70 L documented prior to randomization
* Have an FEV1/FVC ratio <70% documented prior to randomization.
* Have a chest x-ray that is consistent with the diagnosis of COPD and taken <3 months prior to Visit 1. If there is no chest x-ray taken 3 months prior to Visit 1, a chest x-ray will be performed prior to Visit 2.
* Be able to complete all study questionnaires and logs reliably

EXCLUSION CRITERIA: In order to qualify for participation, subjects must not meet any of the following criteria:

* Currently using disallowed medications or will be unable to complete the medication washout periods
* Female subject who is pregnant or lactating
* Have participated in an investigational drug study within 30 days prior to Visit 1 or who is currently participating in another investigational drug study
* Subject whose schedule or travel prevents the completion of all required visits
* Subject who is scheduled for in-patient hospitalization, including elective surgery (in-patient or out-patient) during the trial.
* Subject with life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days prior to Visit 1
* Known history of asthma or any chronic respiratory disease (including a current history of sleep apnea) other than COPD (chronic bronchitis and/or emphysema).
* Subject with a blood eosinophil count >5%
* Subject with clinically significant cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol
* History of cancer except non-melanomatous skin cancer
* History of lung resection of more than one full lobe
* Subject who requires continuous supplemental oxygen therapy. The use of supplemental oxygen, not to exceed 2 L/minute, at nighttime only and/or only during exercise is allowed.
* Have had a change in dose or type of any medications for COPD within 14 days prior to the screening visit
* Have a known sensitivity to (R,R)-formoterol, ipratropium, salmeterol or albuterol or any of the excipients contained in any of these formulations
* Have clinically significant abnormalities that may interfere with the metabolism or excretion of the study drug
* Have a history of substance abuse or drug abuse within 12 months of Visit 1 or with a positive urine drug screen at the screening visit
* Subject with clinically significant abnormal laboratory values
* Subject with clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study
* Subject using any prescription drug for which concomitant beta-agonist administration is contraindicated

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2002-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Overall occurrence of adverse events | Weeks -1, 0, 3, 6, 9, 13, 26, 39, 52

SECONDARY OUTCOMES:
Laboratory parameters | Weeks -1, 0, 3, 6, 9, 13, 26, 39, 52
ECG parameters | Weeks -1, 0, 3, 6, 9, 13, 26, 39, 52
24-hour holter monitoring parameters | Weeks -1, 0, 13, 26, 39, 52
Vital signs | Weeks -1, 0, 3, 6, 9, 13, 26, 39, 52
Plasma arformoterol concentrations | Weeks -1, 0, 3, 6, 9, 13, 26, 39, 52
Physical examination findings | Weeks -1, 53

CONTACTS AND LOCATIONS:
Locations (90):
- United States (90):
  - Pinnacle Research Group, Anniston, Alabama
  - Princeton Pulmonary Group, PC, Birmingham, Alabama
  - Pulmonary & Sleep Associates of Jasper, PC, Jasper, Alabama
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Northern California Research Corp., Fair Oaks, California
  - SARC Research Center, Fresno, California
  - Irvine Center for Clinical Research, Irvine, California
  - Scripps Clinic - Chest and Critical Care, La Jolla, California
  - Torrance Clinical Research, Los Angeles, California
  - Facey Medical Center - Radiant Research, Mission Hills, California
  - Office of Delmer Henninger, MD, Murrieta, California
  - Advanced Clinical Research Institute, Orange, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Advances in Medicine, Rancho Mirage, California
  - Inland Clinical Research, Inc., Riverside, California
  - Institute of Healthcare Assessment, Inc., San Diego, California
  - Wetlin Research Associates, Inc., San Diego, California
  - San Jose Clinical Research, Inc., San Jose, California
  - West Coast Clinical Trials, Signal Hill, California
  - Allergy & Asthma Medical Group of Diablo Valley, Inc., Walnut Creek, California
  - Northern Colorado Pulmonary Consultants, PC, Fort Collins, Colorado
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - University Clinical Research, DeLand, DeLand, Florida
  - nTouch Research, Melbourne, Florida
  - nTouch Research, St. Petersburg, Florida
  - USF Asthma, Allergy and Immunology, Tampa, Florida
  - AHS Medical Research, Inc., Tampa, Florida
  - New Horizon Health Research, Atlanta, Georgia
  - Protocare Trial, Inc., Austell, Georgia
  - nTouch Research, Decatur, Georgia
  - Marietta Pulmonary Medicine, Marietta, Georgia
  - North Point Pulmonary Associates, Roswell, Georgia
  - Pulmonary Consultants, Coeur d'Alene, Idaho
  - University of Chicago - Department of Medicine, Chicago, Illinois
  - Sneeze, Wheeze and Itch, LLC, Normal, Illinois
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Heart of America Research Institute, Shawnee Mission, Kansas
  - Bendel Medical Associates, Lafayette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - North Shore Research Associates, Slidell, Louisiana
  - Office of Paul A. Shapero, MD, PA, Bangor, Maine
  - Primary Care Cardiology Research, Inc., Ayer, Massachusetts
  - Center for Clinical Research, Taunton, Massachusetts
  - ClinSite, Inc., Ann Arbor, Michigan
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Midwest Chest Consultants, PC, Saint Charles, Missouri
  - MedEx HealthCare Research, Inc., St Louis, Missouri
  - C.A.R.E Clinical Research, St Louis, Missouri
  - Office of Keith Popovich, MD, Butte, Montana
  - Montana Medical Research, LLC, Missoula, Montana
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Atlantic Research Associates, Inc., Margate City, New Jersey
  - UrgentMed Family Practice Medical, South Bound Brook, New Jersey
  - Lovelace Scientific Resources - NM, Albuquerque, New Mexico
  - Endwell Family Physicians, Endwell, New York
  - Asthma & Allergy Associates, PC, Ithaca, New York
  - N.Y. Pulmonary Associates, New York, New York
  - Ridgewood Medical Group, Rochester, New York
  - Charlotte Lung and Health Center, Charlotte, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Odyssey Research Services, Fargo, North Dakota
  - Community Research Management Associates, Inc., Cincinnati, Ohio
  - New Horizons Clinical Research, Inc., Cincinnati, Ohio
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Northeast Clinical Research Center, Inc., Allentown, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Consortium Clinical Research, Ltd., Ridley Park, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Spartanburg Pharmaceutical Research, Spartanburg, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Ben Taub General Hospital, Houston, Texas
  - S.W. Asthma Institute, Houston, Texas
  - Breath of Life Research Institute, Houston, Texas
  - Wellmed at Northern Hills, San Antonio, Texas
  - Medsource, Inc., Chesapeake, Virginia
  - Pulmonary Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Commonwealth Clinical Research, Richmond, Virginia
  - Virginia Adult & Pediatric Allergy & Asthma, PC Research Office, Richmond, Virginia
  - Pulmonary Research Partners, Inc., South Boston, Virginia
  - Pulmonary Consultants, PLLC, Tacoma, Washington
  - Morgantown Pulmonary Associates, Morgantown, West Virginia